CLINICAL TRIAL: NCT05295381
Title: Effect of Abdominal Weight Training Assisted by Cough Assist Machine on Lung Function in the Patients With Prolonged Mechanical Ventilation
Brief Title: Abdominal Weight Training Assisted by Cough Assist Machine on Lung Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Shih Feng (Other)
Responsible Party: Sponsor-Investigator, Liu Shih Feng, Chief of department of respiratory therapy in Kaohsiung CGMH, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201900885B0A3
Record Dates: First submitted 2022-02-18; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: PMV
Keywords: prolonged mechanical ventilation; weaning ventilator; abdominal weight training; cough machine

STUDY DESIGN:
Intervention Model Description: AWT group (n=12), AWT+CM group (n=14) control group (n=14).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- abdominal weight training with cough machine (CM) (Experimental): abdominal weight exercise training (sandbag) is maintained for 30 minutes; the starting weight is 1kg to 2kg, and the previous day's weight is maintained each day as well as adding 0.5kg daily. Cough machine training is based on the cough assist machine Comfort Cough II (CC20), in which the inhalation and exhalation times are adjusted to 1-3 seconds, and the positive and negative pressure of the lower pressure 10-15 cmH2O is gradually increased to 30-40 cmH2O for the first time, 4-6 cycles/time, repeated 4-6 times, twice a day, five days a week, until the subject is weaned off the ventilator or transferred out of the ward. A modified Borg scale was used as an indicator of perceived dyspnea.
  Interventions: Device: cough machine (CM); Device: abdominal weight training (AWT)
- abdominal weight training (AWT) without cough machine (CM) (Experimental): abdominal weight exercise training (sandbag) is maintained for 30 minutes; the starting weight is 1kg to 2kg, and the previous day's weight is maintained each day as well as adding 0.5kg daily.
  Interventions: Device: abdominal weight training (AWT)
- control (No Intervention): no abdominal weight training and no cough machine

INTERVENTIONS:
Device: cough machine (CM) — Cough machine training is based on the cough assist machine Comfort Cough II (CC20), in which the inhalation and exhalation times are adjusted to 1-3 seconds, and the positive and negative pressure of the lower pressure 10-15 cmH2O is gradually increased to 30-40 cmH2O for the first time, 4-6 cycles/time, repeated 4-6 times, twice a day, five days a week, until the subject is weaned off the ventilator or transferred out of the ward. A modified Borg scale was used as an indicator of perceived dyspnea.
  Arms: abdominal weight training with cough machine (CM)
Device: abdominal weight training (AWT) — abdominal weight exercise training (sandbag) is maintained for 30 minutes; the starting weight is 1kg to 2kg, and the previous day's weight is maintained each day as well as adding 0.5kg daily.
  Arms: abdominal weight training (AWT) without cough machine (CM); abdominal weight training with cough machine (CM)

SUMMARY:
The patients with prolonged mechanical ventilation (PMV) have the risk of ineffective coughing and infection due to diaphragm weakness, making it more difficult to wean. This study aimed to explore the intervention of abdominal weight training (AWT) with/ without cough machine (CM) on lung function, respiratory muscle strength and cough ability in these patients.

DETAILED DESCRIPTION:
Methods 40 patients with PMV were randomly assigned to three groups: AWT group (n=12), AWT+CM group (n=14) and control group (n=14). The effectiveness on pulmonary function, respiratory muscle strength and cough ability were compared among these three groups.

ELIGIBILITY:
Inclusion Criteria:

* (1) Invasive ventilator users,
* (2) Hemodynamically stable,
* (3) Intubated endotracheal tube or tracheotomy tube,
* (4) Clearly conscious and cooperative,
* (5) Vital capacity (VC) <10ml/kg

Exclusion Criteria:

* (1) Unconscious or unwilling to sign the informed consent form,
* (2) No spontaneous breathing,
* (3) Active bleeding with unstable hemodynamics,
* (4) Acute infection symptoms,
* (5) Abdominal distension, digestion problems (including nausea and vomiting),
* (6) Severe heart failure (ejection fraction ≤ 30%),
* (7) Unhealed wounds in the chest and abdomen,
* (8) Bullous emphysema,
* (9) Sensitive pneumothorax or mediastinal pneumothorax,
* (10) Recent history of traumatic stress,
* (11) Acute head and neck injury (unless the injury site is immobilized)

Ages: 57 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Maximum inspiratory pressure change by the intervention | Change between 1 day before and 2 weeks after the intervention
  lung function
Maximum expiratory pressure change by the intervention | Change between 1 day before and 2 weeks after the intervention
  lung function

SECONDARY OUTCOMES:
vital capacity change by the intervention | Change between 1 day before and 2 weeks after the intervention
  lung function

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Tang Hsieh, Study Chair — Institutional Review Board Chang Gung Medical Foundation
Locations (1):
- Chang Gung Medical Foundation, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim SM, Choi WA, Won YH, Kang SW. A Comparison of Cough Assistance Techniques in Patients with Respiratory Muscle Weakness. Yonsei Med J. 2016 Nov;57(6):1488-93. doi: 10.3349/ymj.2016.57.6.1488. PMID 27593879
- [Result] Lacombe M, Del Amo Castrillo L, Bore A, Chapeau D, Horvat E, Vaugier I, Lejaille M, Orlikowski D, Prigent H, Lofaso F. Comparison of three cough-augmentation techniques in neuromuscular patients: mechanical insufflation combined with manually assisted cough, insufflation-exsufflation alone and insufflation-exsufflation combined with manually assisted cough. Respiration. 2014;88(3):215-22. doi: 10.1159/000364911. Epub 2014 Aug 21. PMID 25171575
- [Result] Sivasothy P, Brown L, Smith IE, Shneerson JM. Effect of manually assisted cough and mechanical insufflation on cough flow of normal subjects, patients with chronic obstructive pulmonary disease (COPD), and patients with respiratory muscle weakness. Thorax. 2001 Jun;56(6):438-44. doi: 10.1136/thorax.56.6.438. PMID 11359958
- [Derived] Hung TY, Wu WL, Kuo HC, Liu SF, Chang CL, Chang HC, Tsai YC, Liu JF. Effect of abdominal weight training with and without cough machine assistance on lung function in the patients with prolonged mechanical ventilation: a randomized trial. Crit Care. 2022 May 25;26(1):153. doi: 10.1186/s13054-022-04012-1. PMID 35614518